CLINICAL TRIAL: NCT01449487
Title: A Randomized, Double-blind, Cross-over Trial in Patients With Irritable Bowel Syndrome Investigating the Efficacy and Safety of PPC-5650 on Sensation and Pain During Standardized Stimulation of the Rectosigmoid
Brief Title: Investigation of Efficacy and Safety of PPC-5650 to Experimental Induced Sensation and Pain in the Rectosigmoid
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Aros Pharma ApS (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: Aros-001
Record Dates: First submitted 2011-09-30; First posted 2011-10-10 (Estimated); Last update posted 2014-05-21 (Estimated); Status verified 2014-05

CONDITIONS: Pain
Keywords: Experimental pain; IBS; Rectum
MeSH Terms: conditions — Pain

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- PPC-5650 (Active Comparator)
  Interventions: Drug: PPC-5650
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: PPC-5650 — Solution for administration in the rectum Single dose of 25µg/ml at a volume of 50ml
  Other Names: No other name
  Arms: PPC-5650
Drug: Placebo — Solution for administration in the rectum Identical tp active solution but without active drug
  Other Names: No other name
  Arms: Placebo

SUMMARY:
Irritable Bowel Syndrome (IBS) is a gastrointestinal disorder characterized by chronic abdominal pain and altered bowel habits in the absence of any organic cause. Patients with IBS visit the doctor more frequently, use more diagnostic tests, consume more medications, miss more workdays, and consume more overall direct costs than patients without IBS. More specific treatment of the localized symptoms of IBS is therefore needed, why the present study will investigate the effect and mechanisms of PPC-5650. PPC-5650 is a new chemical entity that can negatively modulate the activity of Acid sensing ion channels (ASICs). It is a potent low molecular weight inhibitor for this class of ion channels described to date.

It is hypothesized that safety, efficacy and mechanisms of local administration in the rectum of PPC-5650 can be evaluated by use of experimental induced sensation and pain in the rectum.

DETAILED DESCRIPTION:
Clinical pain and especially visceral pain is diffuse and widespread, and normally associated with many autonomic symptoms that may blur the characterization of disease in clinical practice. When treating clinical pain analgesic effects are difficult to evaluate due to a number of factors other than the pain intensity. These modifiers of the effect may include complaints relating to psychological, cognitive and social aspects of the illness, as well as systemic reactions. Hence, any change in these factors will invariably also interfere with pain intensity and pain quality and bias the assessment of analgesics in clinical trials.

Because of the confounders mentioned above, experimental pain models are often advantageous for characterizing analgesics. Basic mechanisms in pain perception, transduction and central processing can also be explored by means of human experimental pain models. These models, when applied to healthy volunteers or to patients, provide an important translational link between preclinical animal testing and human clinical trials. In clear contrast to clinical pain, experimental pain models allow the possibility of controlling the duration, the intensity and the nature of the pain stimulus. As pain is a multidimensional perception it is obvious that the reaction to a single stimulus of a certain modality only represents a limited part of the pain experience and therefore a variety of stimulus modalities are required to mimic the clinical situation. By use of a multi-modal pain model it is possible to induce sensation and pain in the rectum, investigating safety, effect and mechanisms of drugs.

This is an exploratory study investigating effect, mechanisms and safety of PPC-5650 to experimental induced pain in patients with IBS. The study aims to provide data to support further evaluation of PPC-5650 in the gastrointestinal area.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent
* Postmenopausal women or women who have undergone hysterectomy, and males between 18 and 70 years of age
* Pain intensity during pain attack should be >5 on the GSRS questionnaire
* Hypersensitivity within the last 2 years measured with the barostat
* Patients able to co-operate and tolerate the experimental procedures (as assessed in the training visit)
* Patients on stable medication
* Only patients that do not take over the counter medication 24h before the two study sessions

Exclusion Criteria:

* Any history of, or current condition or medication that, as judged by the investigator, may affect gastrointestinal function and the interpretation of the clinical data
* Any clinically relevant abnormal values from the laboratory tests on hematology, clinical chemistry, urine analyses and/or faeces testing, as judged by the investigator.
* Chronic extraintestinal pain dominating the clinical history
* Any known biochemical or structural abnormality of the digestive tract such as gluten enteropathy, bile acid diarrhea, lymphocytic colitis and/or collagenous colitis, Chronic inflammatory bowel diseases, chronic pancreatitis
* Major intra-abdominal surgery; appendectomy and minor laparoscopic gynecological surgery acceptable.
* Any planned surgical intervention within the duration of the trial.
* Any abdominal surgery
* Participation in any other clinical trial within three months prior to the pre-screening visit.
* Alcohol or drug abuse.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2012-01; Primary Completion 2013-05 (Actual); Study Completion 2013-05 (Actual)

PRIMARY OUTCOMES:
Effect of PPC-5650 | Change in pain from baseline to 120 minutes
  Outcome measurements are achieved by use of multimodal pain responses (thermal, mechanical, electrical) in the rectosigmoid.

SECONDARY OUTCOMES:
Safety profile of PPC-5650 | Change from baseline to 120 minutes
  By recording adverse effects as well as fysiological characters e.g. blood pressure, pulse, ECG is will be possible to assess safety profile of PPC-5650
Effect of PPC-5650 | Change in pain from baseline to 120 minutes
  Outcome is achieved by measuring pain and sensory responses to experimental induced pain in the rectosigmoid by use of visual analogue scale (VAS) at VAS=1, 3, 5 and 7
Central mechanisms | Change from baseline to 120 minutes
  This outcome is done by use of referred pain areas to the experimental induced pain in the rectosigmoid
Objective pain | Change from baseline to 120 minutes
  Assessment of objective pain will be done by recording evoked brain potentials to electrical stimulation in the rectosigmoid

CONTACTS AND LOCATIONS:
Overall Officials: Asbjørn M Drewes, Professor, Study Director — Mech-Sense, Aalborg Hospital, Aalborg, Denmark
Locations (1):
- Department of Gastroenterology, Gothenburg, Sweden

REFERENCES:
- See also: Information regarding multi-modal probe used for inducing experimental pain in the rectum — http://www.mech-sense.com